CLINICAL TRIAL: NCT07340775
Title: Hypersensitivity to Amylin in Post-Traumatic Headache: A Randomized Clinical Trial
Brief Title: Hypersensitivity to Amylin in Post-Traumatic Headache
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Ksenija Cucanic, PhD Fellow, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-21067689
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Headache Disorders, Secondary; Brain Diseases; Headache Disorders; Nervous System Diseases; Central Nervous System Diseases; Neurologic Manifestations; Signs and Symptoms; Pathological Conditions, Signs and Symptoms; Post-Traumatic Headache; Pain; Peptide Hormones; Hormones; Hormones, Hormone Substitutes, and Hormone Antagonists; Peptides; Amino Acids, Peptides, and Proteins; Amylin; Pramlintide
Keywords: Post-traumatic headache; Pain; Amylin
MeSH Terms: conditions — Headache Disorders, Secondary; Brain Diseases; Headache Disorders; Nervous System Diseases; Central Nervous System Diseases; Neurologic Manifestations; Signs and Symptoms; Pathological Conditions, Signs and Symptoms; Post-Traumatic Headache; Pain | interventions — Islet Amyloid Polypeptide

STUDY DESIGN:
Intervention Model Description: This single-center trial applies a randomized, double-blind, placebo-controlled, two-way crossover design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amylin (Experimental): Pramlintide (Amylin) will be administered by intravenous infusion.
  Interventions: Drug: Amylin
- Placebo (Placebo Comparator): Placebo (isotonic saline) will be administered by intravenous infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amylin — The participants will receive continuous intravenous infusion of 6 μg/min of pramlintide (amylin) over 20 minutes.
  Arms: Amylin
Drug: Placebo — The participants will receive continuous intravenous infusion of 20 mL of placebo (isotonic saline) over 20 minutes.
  Arms: Placebo

SUMMARY:
Pramlintide is a peptide analogue of human amylin which is a vasoactive substance involved in the pathogenesis of headache. This study investigates whether pramlintide induces migraine-like headache in people with persistent post-traumatic headache (PTH) attributed to mild traumatic brain injury (mTBI).

DETAILED DESCRIPTION:
Amylin is a vasodilator released from nerve fibers within the trigeminovascular system, which is considered a key anatomical and physiological substrate in the pathogenesis of migraine and persistent post-traumatic headache (PTH). Persistent PTH attributed to mild traumatic brain injury frequently presents with migraine attacks, suggesting shared underlying mechanisms with migraine. This study aims to determine whether intravenous infusion of pramlintide, an analogue of amylin, can induce migraine-like headache in individuals with persistent post-traumatic headache. To test this hypothesis, we will conduct a randomized, double-blind, placebo-controlled, two-way crossover study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years of age upon entry into screening
* History of persistent headache attributed to mild traumatic injury to the head for ≥ 12 months and in accordance with the International Classification of Headache Disorders, 3rd Edition (ICHD-3)
* ≥ 4 monthly headache days on average across the 3 months prior to screening
* Provision of informed consent prior to initiation of any study-specific activities/procedures

Exclusion Criteria:

* > 1 mild traumatic injury to the head
* History of any primary or secondary headache disorder prior to mild traumatic injury to the head (except for infrequent episodic tension-type headache)
* History of moderate or severe injury to the head
* History of whiplash injury
* History of craniotomy
* History or evidence of any other clinically significant disorder, condition or disease (except for those outlined above) than, in the opinion of the site investigator, would pose a risk to subject safety or interfere with study evaluation, procedures or completion
* The subject is at risk of self-harm or harm to others as evidenced by past suicidal behavior
* Female subjects of childbearing potential with a positive pregnancy test during any study visit
* Cardiovascular disease of any kind, including cerebrovascular diseases
* Hypertension (systolic blood pressure of ≥150 mmHg and/or diastolic blood pressure of ≥100 mmHg) prior to the start of infusion on the experimental day
* Hypotension (systolic blood pressure of ≤90 mmHg and/or diastolic blood pressure of ≤50 mmHg)
* Initiation, discontinuation, or change of dosing of prophylactic medications within 2 months prior to study inclusion
* Intake of acute medications (e.g. analgesics, triptans) within 48 hours of infusion start
* Baseline headache intensity of >3 on an 11-point numeric rating scale (0 being no headache, 10 being the worst imaginable headache)
* Baseline migraine-like headache or self-reported baseline headache that mimics the subjects' usual migraine-like headache

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of migraine-like headache | 12 hours
  Difference in incidence of migraine-like headache (0 to 12 hours) between pramlintide and placebo.

SECONDARY OUTCOMES:
Headache Intensity Scores | 12 hours
  Difference in area under the curve (AUC) for headache intensity scores (0 to 12 hours) between pramlintide and placebo.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Access Criteria: Anonymized data not published within this article will be made available on reasonable request from any qualified investigator.

REFERENCES:
- [Background] Asmar M, Bache M, Knop FK, Madsbad S, Holst JJ. Do the actions of glucagon-like peptide-1 on gastric emptying, appetite, and food intake involve release of amylin in humans? J Clin Endocrinol Metab. 2010 May;95(5):2367-75. doi: 10.1210/jc.2009-2133. Epub 2010 Mar 1. PMID 20194711
- [Background] Hay DL, Chen S, Lutz TA, Parkes DG, Roth JD. Amylin: Pharmacology, Physiology, and Clinical Potential. Pharmacol Rev. 2015 Jul;67(3):564-600. doi: 10.1124/pr.115.010629. PMID 26071095
- [Background] Ghanizada H, Al-Karagholi MA, Walker CS, Arngrim N, Rees T, Petersen J, Siow A, Morch-Rasmussen M, Tan S, O'Carroll SJ, Harris P, Skovgaard LT, Jorgensen NR, Brimble M, Waite JS, Rea BJ, Sowers LP, Russo AF, Hay DL, Ashina M. Amylin Analog Pramlintide Induces Migraine-like Attacks in Patients. Ann Neurol. 2021 Jun;89(6):1157-1171. doi: 10.1002/ana.26072. Epub 2021 Apr 8. PMID 33772845
- [Background] Ashina H, Porreca F, Anderson T, Amin FM, Ashina M, Schytz HW, Dodick DW. Post-traumatic headache: epidemiology and pathophysiological insights. Nat Rev Neurol. 2019 Oct;15(10):607-617. doi: 10.1038/s41582-019-0243-8. Epub 2019 Sep 16. PMID 31527806
- [Background] Ashina H, Iljazi A, Al-Khazali HM, Ashina S, Jensen RH, Amin FM, Ashina M, Schytz HW. Persistent post-traumatic headache attributed to mild traumatic brain injury: Deep phenotyping and treatment patterns. Cephalalgia. 2020 May;40(6):554-564. doi: 10.1177/0333102420909865. Epub 2020 Feb 26. PMID 32102546
- [Background] Rasmussen BK, Olesen J. Symptomatic and nonsymptomatic headaches in a general population. Neurology. 1992 Jun;42(6):1225-31. doi: 10.1212/wnl.42.6.1225. PMID 1603351
- [Background] Ashina H, Eigenbrodt AK, Seifert T, Sinclair AJ, Scher AI, Schytz HW, Lee MJ, De Icco R, Finkel AG, Ashina M. Post-traumatic headache attributed to traumatic brain injury: classification, clinical characteristics, and treatment. Lancet Neurol. 2021 Jun;20(6):460-469. doi: 10.1016/S1474-4422(21)00094-6. PMID 34022171
- See also: Related Info — https://www.regionh.dk/til-fagfolk/forskning-og-innovation/de-regionale-videnskabsetiske-komiteer/sider/default.aspx